CLINICAL TRIAL: NCT06750887
Title: Modifying Lumbar Flexion Pain Thresholds in Patients With Chronic Low Back Pain Through Visual-proprioceptive Manipulation With Virtual Reality: a Cross-sectional Study
Brief Title: Modifying Lumbar Flexion Pain Thresholds in Chronic LBP Using Virtual Reality and Visual-Proprioceptive Manipulation
Acronym: CLEVER-BODY
Status: Completed | Type: Observational
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Chair Profesor, Cardenal Herrera University
Other Study IDs: Cardenal Herrera University 70; PID2020-115609RB-C22 (Other Grant/Funding Number: MINISTRY OF SCIENCE AND INNOVATION OF SPAIN)
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Chronic Low Back Pain (CLBP)
Keywords: chronic low back pain; virtual reality; flexion-evoked pain; illusions; central processing
MeSH Terms: conditions — Illusions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- NORMAL CONDITION: The normal condition is measured as a lumbar flexion without VR until the onset of pain.
  Interventions: Other: Normal condition
- UNDERSTATED CONDITION: It involves an illusion with virtual reality where the patients perform a lumbar flexion until the onset of pain and they feel a 20% less movement in the VR (understated visual feedback)
  Interventions: Other: Understated condition
- OVERSTATED CONDITION: It involves an illusion with virtual reality where the patients perform a lumbar flexion until the onset of pain and they feel a 20% more movement in the VR (understated visual feedback)
  Interventions: Other: OVERSTATED CONDITION

INTERVENTIONS:
Other: Normal condition — The normal condition IS measured as a lumbar extension without VR until the onset of pain.
  Groups: NORMAL CONDITION
Other: Understated condition — It involves an illusion with virtual reality where the patients perform a lumbar flexion until the onset of pain and they feel a 20% less movement in the VR (understated visual feedback)
  Groups: UNDERSTATED CONDITION
Other: OVERSTATED CONDITION — It involves an illusion with virtual reality where the patients perform a lumbar flexion until the onset of pain and they feel a 20% more movement in the VR (understated visual feedback)
  Groups: OVERSTATED CONDITION

SUMMARY:
This study investigates the potential to modify movement-evoked pain in individuals with chronic low back pain (LBP) by manipulating visual proprioceptive feedback through virtual reality (VR). Fifty patients with non-specific chronic LBP are planned to participate. Participants perform lumbar spine flexions until pain onset under three conditions: accurate visual feedback (control), feedback showing 20% less movement (F-), and feedback showing 20% more movement (F+). Lumbar range of motion (ROM) is measured using a 3-space Fastrack motion analysis system. The study also explores whether individuals with higher pain levels, kinesiophobia, or catastrophising are more susceptible to VR feedback manipulation. Pain thresholds, pain intensity, kinesiophobia, and catastrophising levels are assessed.

DETAILED DESCRIPTION:
This study investigates the potential to modify movement-evoked pain in individuals with chronic low back pain (LBP) by manipulating visual proprioceptive feedback through virtual reality (VR). The research aims to explore how altering the perception of movement through VR can influence pain experiences and motor behavior. A total of 50 patients with non-specific chronic LBP are planned to participate.

Participants will perform lumbar spine flexion movements until the onset of pain under three experimental conditions: (1) accurate visual feedback, without virtual reality (control); (2) underestimated movement feedback (F-), where the VR displays 20% less movement than performed; and (3) overestimated movement feedback (F+), where the VR shows 20% more movement than actually executed. These conditions are designed to evaluate how changes in visual feedback impact pain perception and range of motion (ROM).

Lumbar ROM will be objectively measured using a 3-space Fastrack motion analysis system to ensure precise tracking of movement. The study also seeks to identify whether individuals with higher levels of pain, kinesiophobia (fear of movement), or catastrophising (an exaggerated negative mindset about pain) are more susceptible to VR feedback manipulation.

Various psychological and physical metrics will be assessed using validated tools, including pain thresholds, pain intensity, kinesiophobia, and catastrophising levels. This comprehensive approach aims to identify patient subgroups who may benefit most from VR-based interventions and to shed light on the mechanisms by which altered visual feedback modifies pain perception and motor behavior in chronic LBP.

ELIGIBILITY:
Inclusion Criteria:

* Participants of both sexes.
* Aged between 18 and 65 years.
* Diagnosed with non-specific chronic low back pain (according to the European COST B13 guidelines).
* Presence of lumbar extension limitation.

Exclusion Criteria:

* Diagnosis of a spinal tumor.
* Presence of a spinal infection or fracture.
* Diagnosed systemic diseases.
* Diagnosis of fibromyalgia.
* Presence of cauda equina syndrome.
* History of prior spinal surgery.
* Musculoskeletal injuries of the lower extremities (including: sciatica; radiating pain in the lower extremities; symptoms of numbness or weakness in the lower extremities)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic low back pain
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-12-04 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
MOVEMENT EVOKED PAIN THRESHOLD | Baseline (pre-intervention) and immediately post-intervention (at 50 minutes)
  The maximum lumbar ROM without pain was measured in each condition using a 3-Space Fastrack motion analysis system.
Pain Interference and Pain Intensity | Baseline (pre-intervention) and immediately post-intervention (at 50 minutes)
  The Brief Pain Inventory (BPI) is a pain assessment tool designed to measure pain intensity and interference with daily functioning in patients with low back pain
Fear of movement | Baseline (pre-intervention) and immediately post-intervention (at 50 minutes)
  We will use the reliable and validated Spanish version of the Tampa Scale for Kinesiophobia (TSK), which consists of 11 independent phrases rated on a 4-point scale (1 = totally disagree to 4 = totally agree). Higher scores indicate higher levels of fear of movement.

SECONDARY OUTCOMES:
Catastrophizing | Baseline (pre-intervention) and immediately post-intervention (at 50 minutes)
  The validated Spanish version of the Pain Catastrophizing Scale (PCS) will be applied, which has demonstrated internal consistency, test-retest reliability, and sensitivity to change. The PCS comprises 13 items rated on a 5-point scale from 0 (never) to 4 (always) that measure 3 components of catastrophising: rumination, magnification, and helplessness. Higher scores indicate greater pain-related catastrophising.

CONTACTS AND LOCATIONS:
Locations (1):
- Arnau de Vilanova Hospital, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Harvie DS, Broecker M, Smith RT, Meulders A, Madden VJ, Moseley GL. Bogus visual feedback alters onset of movement-evoked pain in people with neck pain. Psychol Sci. 2015 Apr;26(4):385-92. doi: 10.1177/0956797614563339. Epub 2015 Feb 17. PMID 25691362
- [Derived] Jordan-Lopez J, Arguisuelas MD, Domenech J, Penalver-Barrios ML, Miragall M, Herrero R, Banos RM, Amer-Cuenca JJ, Lison JF. Modifying lumbar flexion pain thresholds in patients with chronic low back pain through visual-proprioceptive manipulation with virtual reality: a cross-sectional study. J Neuroeng Rehabil. 2025 Jun 19;22(1):138. doi: 10.1186/s12984-025-01664-2. PMID 40537791